CLINICAL TRIAL: NCT00004940
Title: Phase III Study of L-Cysteine in Patients With Erythropoietic Protoporphyria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13376; BWH-FDR000996-DR
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Erythropoietic Protoporphyria
Keywords: erythropoietic protoporphyria; inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Metabolism, Inborn Errors; Porphyrias; Rare Diseases | interventions — Cysteine

INTERVENTIONS:
Drug: cysteine hydrochloride

SUMMARY:
OBJECTIVES:

I. Determine the long-term efficacy and safety of L-cysteine in the prevention photosensitivity in patients with erythropoietic protoporphyria.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a phase III study, lasting 3 years; 1996-1999. Patients are administered L-cysteine orally twice daily, 2 capsules with breakfast and 2 with lunch.

Patients fill in questionnaires and diary sheets about their reaction to sunlight exposure, and have blood tested 3 times a year.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Erythropoietic protoporphyria RBC protoporphyrin greater than 50 micrograms/100 dL

--Prior/Concurrent Therapy--

At least 3 months since prior betacarotene or L-cysteine

No concurrent betacarotene

--Patient Characteristics--

* Fertile female patients must use effective contraception for duration of trial and for 3 weeks thereafter
* Not pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1996-05; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Micheline Mary Mathews-Roth, Study Chair — Brigham and Women's Hospital